CLINICAL TRIAL: NCT04608136
Title: Egg Yolk and Underlying Metabolisms on Modifying HDL Levels and Associated Genetics in Individuals With Metabolic Syndrome
Brief Title: Egg Yolk and Underlying Metabolisms on Modifying HDL Levels in Individuals With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: National Research Council of Thailand (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MU-CIRB 2019/255.0310
Record Dates: First submitted 2020-09-21; First posted 2020-10-29 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Metabolic Syndrome
Keywords: metabolic syndrome; diabetes; diet; eggs; cholesterol; weight loss
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yolk ketogenic diet (Experimental): consume carbohydrate < 10% and 3 whole eggs supplement per day in 12 weeks
  Interventions: Behavioral: Diet intervention
- White ketogenic diet (Experimental): consume carbohydrate < 10% and 6 white eggs supplement per day in 12 weeks
  Interventions: Behavioral: Diet intervention
- Control group (Active Comparator): decrease consumption of diet from typical (decreased energy 20%) but consume carbohydrate in normal level
  Interventions: Behavioral: Diet intervention

INTERVENTIONS:
Behavioral: Diet intervention — Volunteers will be instructed on dietary recommendation throughout the research program to achieve a stable daily energy intake.

SUMMARY:
This research compare the effects of low carbohydrate intake and consumption of 3 eggs per day, and low energy diet on diabetes control and biomarkers of CVD in obese people.

DETAILED DESCRIPTION:
This research study examines the effects of changes in weight, metabolism of glucose and cholesterol in the blood through diet and behavior modification. The main objective of this study was to compare the effects of low carbohydrate intake and consumption of 3 eggs per day, and low energy diet on diabetes control and biomarkers of CVD in obese people. In addition, HDL quantity and size as well as HDL function was compared between the group who ate the whole egg and the group who did not eat the yolk.

ELIGIBILITY:
Inclusion Criteria:

1. weight stable > 3 months (changing < 5%)
2. three or more of the following five criteria are met 2.1 waist circumference ≥ 90 cm (men) or ≥ 80 cm (women) 2.2 fasting blood sugar ≥ 100 mg/dl 2.3 fasting triglyceride (TG) level ≥ 150 mg/dl 2.4 fasting high-density lipoprotein (HDL) cholesterol level ≤ 40 mg/dl (men) or ≤ 50 mg/dl (women) 2.5 blood pressure over 130/85 mmHg
3. can consume food that provided in project
4. healthy

Exclusion Criteria:

1. consume drugs i.e. weight loss drugs, herbal pills, asthma drugs, steroid drugs, thyroid drugs, insulin injections, SGLT1 inhibitors drugs, SGLT2 inhibitors drugs, sulfonylurea drugs, blood lipid-lowering drugs
2. people who exercise vigorously (> 150 minutes per week)
3. people who are or have weight loss by consuming less than 30% of carbohydrates, or are losing weight by other methods or who have eaten a specific diet as prescribed by a doctor within the past 6 months
4. people who drink alcohol more than once a week
5. people who had a LDL level within 6 months > 190 mg/dl
6. fasting blood glucose levels > 250 mg/dl and using diabetes drugs other than metformin
7. people with heart disease, type 1 diabetes, renal impairment > level 3A
8. history of cancer, lung disease, gastrointestinal disease
9. people who smoke, people with eating disorder, people who have received psychiatric drugs
10. become a volunteer in a research project that is conducting a study related to food consumption
11. people who are unable to keep up with the treatment or are expected to be absent in this area for the next 4 months
12. pregnancy or breastfeeding
13. egg allergy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Changes in weight following dietary intervention | Baseline and after 12 weeks
  weight (kg) analysis
Changes in body mass index following dietary intervention | Baseline and after 12 weeks
  body mass index (kg/m^2) analysis
Changes in waist circumference following dietary intervention | Baseline and after 12 weeks
  waist circumference (cm) analysis
Changes in lipid profiles concentration following dietary intervention | Baseline and after 12 weeks
  Triglycerides (mg/dl), Cholesterol (mg/dl), HDL-cholesterol (mg/dl) and LDL-cholesterol (mg/dl) concentration analysis
Changes in blood glucose and insulin concentration following dietary intervention | Baseline and after 12 weeks
  HbA1C (%), glucose (mg/dl) and insulin (mg/dl) concentration analysis
Changes in betahydroxybutirate concentration following dietary intervention | Baseline and after 12 weeks
  betahydroxybutirate (mmol/L) concentration analysis
Changes in electrolytes concentration following dietary intervention | Baseline and after 12 weeks
  Na+ (mg/dl), K+ (mg/dl), Cl- (mg/dl) and HCO3- (mg/dl) concentration analysis
Changes in physical activity | Baseline and after 12 weeks
  physical activity (MET-minutes/week) collect data by using questionnaires
Change from baseline Glycemia at 180 minutes | Minutes after intake of 75 g glucose: 0, 30, 60, 90, 120, 180
  glucose (mg/dl)
Change from baseline Insulin at 180 minutes | Minutes after intake of 75 g glucose: 0, 30, 60, 90, 120, 180
  insulin (μU/ml)

SECONDARY OUTCOMES:
Changes in blood pressure | Baseline and after 12 weeks
  systolic and diastolic blood pressure (mmHg)
Changes in fasting leptin levels | Baseline and after 12 weeks
  leptin (mg/dl) concentration analysis
Changes in energy intake following dietary intervention | Baseline and after 12 weeks
  energy (kcal)
Changes in carbohydrate following dietary intervention | Baseline and after 12 weeks
  carbohydrate (g)
Changes in protein intake following dietary intervention | Baseline and after 12 weeks
  protein (g)
Changes in fat intake following dietary intervention | Baseline and after 12 weeks
  fat (g)

CONTACTS AND LOCATIONS:
Overall Officials: Korapat Mayurasakorn, MD., Principal Investigator — Doctor in Family Medicine
Locations (1):
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok Noi, Bangkok, Thailand

REFERENCES:
- [Derived] Pinsawas B, Surawit A, Mongkolsucharitkul P, Pongkunakorn T, Suta S, Manosan T, Ophakas S, Pumeiam S, Sranacharoenpong K, Mayurasakorn K. Asian Low-Carbohydrate Diet with Increased Whole Egg Consumption Improves Metabolic Outcomes in Metabolic Syndrome: A 52-Week Intervention Study. J Nutr. 2024 Nov;154(11):3331-3345. doi: 10.1016/j.tjnut.2024.08.027. Epub 2024 Sep 7. PMID 39245182